CLINICAL TRIAL: NCT07073872
Title: The Effect of Nurse-Led Discharge Education Based on IDEAL Discharge Planning on Discharge Satisfaction and Readmission Rates in Laparoscopic Abdominal Surgery Patients
Brief Title: IDEAL Discharge Education Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Collaborators: Kutahya Health Sciences University (Other); Anadolu Medical Center (Other)
Responsible Party: Principal Investigator, Gizemnur Torun, Principal Inversigator, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ASM-EK-24/259
Record Dates: First submitted 2025-06-27; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Laparoscopic Abdominal Surgeries
Keywords: discharge education; IDEAL discharge; teach-back; nurse-led
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IDEAL Discharge Education Program (IDEP) (Experimental): IDEAL Discharge Education Program (IDEP)
  Interventions: Other: IDEAL Discharge Education Program
- Control Group (Active Comparator): control group
  Interventions: Other: control group

INTERVENTIONS:
Other: IDEAL Discharge Education Program — Participants in the intervention group received the nurse-led IDEAL Discharge Education Program (IDEP) and the control group received a standard 15-minute face-to-face discharge education the day of discharge day. The IDEP is a nurse-led, structured discharge education program in accordance with IDEAL Discharge Planning that uses the teach-back method. IDEP is an individualized discharge educational program for surgical patients that utilizes the teach-back method and a printed booklet.
  Arms: IDEAL Discharge Education Program (IDEP)
Other: control group — This group receives routine hospital discharge instructions for 15 minutes on the day of discharge.
  Arms: Control Group

SUMMARY:
Background: Patients after laparoscopic abdominal surgery are frequently seen with complications such as pain and infection after discharge, which affects the readmission rate of patients to hospital. It is predicted that these complications will be reduced with IDEAL (Include, Discuss, Educate, Assess, and Listen) discharge education given during discharge and patient satisfaction will increase.

Objectives: The aim of this quasi-experimental study was to investigate the effect of discharge education prepared in accordance with IDEAL discharge planning recommendations on discharge satisfaction levels and readmission rates in laparoscopy abdominal surgery patients.

Methods: Patients were recruited from an internationally accredited hospital in Kocaeli, Turkey between February and August 2024. This study was conducted on 62 patients (31 in each intervention and control group). Participants in the intervention group received the nurse-led IDEAL Discharge Education Program (IDEP) and the control group received a standard 15-minute face-to-face discharge education the day of discharge day. The IDEP is a nurse-led, structured discharge education program in accordance with IDEAL Discharge Planning that uses the teach-back method. IDEP is an individualized discharge educational program for surgical patients that utilizes the teach-back method and a printed booklet. Data on discharge education satisfaction was measured at day of discharge (T1), and rehospitalization and readmission was assessed at 1-month after discharge (T2). Outcomes were analyzed with Independent Samples t Test and Chi Square.

ELIGIBILITY:
Inclusion Criteria:

* Undergone laparoscopic abdominal surgery
* Be hospitalized for at least 24 hours
* Speak and understand Turkish
* Be 18 years of age or older

Exclusion Criteria:

* Have undergone revision surgery
* Patients with communication difficulties due to any medical condition
* Patients who refused to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2024-09-08 (Actual)

PRIMARY OUTCOMES:
Discharge Education Satisfaction Scale for Surgical Patients | Day 1
  Satisfaction with the discharge education program was assessed using the Discharge Education Satisfaction Scale for Surgical Patients. The scale's scores range from a minimum of 21 to a maximum of 105, with higher scores reflecting greater satisfaction.
Readmission rate | 1st month
  Readmission rate
Rehospitalization rate | 1st month
  Rehospitalization rate

CONTACTS AND LOCATIONS:
Locations (1):
- Anadolu Medical Center, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No